CLINICAL TRIAL: NCT04459039
Title: Do We Need Fluid Restriction After Stapled Hemorrhoidopexy? A Pilot, Double-Blinded, Randomized Controlled Trial
Brief Title: Fluid Restriction After Stapled Hemorrhoidopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chiao Cheng, Division of Colon and Rectal Surgery, Department of Surgery, Tri-Service General Hospital, National Defense Medical Center, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2-106-05-063
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Fluid Restriction
Keywords: Stapled hemorrhoidopexy; Fluid restriction; Urinary retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluid restriction (Experimental): Within 12 h of surgery, the experimental group received 1000 mL 0.9% sterile saline intravenously.
  Interventions: Drug: 1000 mL 0.9% sterile saline
- Non-fluid restriction (Placebo Comparator): Within 12 h of surgery, the control group received 250 mL 0.9% sterile saline intravenously
  Interventions: Drug: 250 mL 0.9% sterile saline

INTERVENTIONS:
Drug: 1000 mL 0.9% sterile saline — Within 12 h of surgery, the experimental group received 1000 mL 0.9% sterile saline intravenously.
  Arms: Fluid restriction
Drug: 250 mL 0.9% sterile saline — Within 12 h of surgery, the control group received 250 mL 0.9% sterile saline intravenously.
  Arms: Non-fluid restriction

SUMMARY:
BACKGROUND: Conventional hemorrhoidectomy leads to a high urinary retention rate and fluid restriction is commonly recommended to minimize complications. However, the need for postoperative fluid restriction among patients who have undergone stapled hemorrhoidopexy is unclear. We aimed to determine whether fluid restriction after stapled hemorrhoidopexy with/without partial external hemorrhoidectomy could reduce urinary retention and postoperative pain.

PATIENTS AND METHODS: In this prospective, double-blinded, randomized controlled trial, we enrolled patients who had grade III or IV hemorrhoids and underwent stapled hemorrhoidopexy with/without partial external hemorrhoidectomy; 250 mL/12 h of sterile 0.9% saline was administered to the fluid restriction group after the operation, and 1000 mL/12 h was given to the non-fluid-restriction group. We focused on the need for fluid restriction after stapled hemorrhoidopexy.

ELIGIBILITY:
Inclusion Criteria:

* Gr. III-IV hemorrhoids paitents

Exclusion Criteria:

* Age<20 or >80
* Allergy to NSAID or opoids
* Impaired renal function
* Pregnant or breast feeding

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
first urination | 1 day
  the time to first urination after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan